CLINICAL TRIAL: NCT04800419
Title: Randomized Controlled Trial of Mindfulness-based Stress Reduction in Newly Diagnosed Head and Neck Cancer: Assessing Their Effect on Positive Psychology and Quality of Life
Brief Title: RCT of Effects of Mindfulness-based Stress Reduction in Head and Neck Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universiti Sains Malaysia (Other)
Collaborators: Henan Medical University (Other)
Responsible Party: Principal Investigator, Mohammad Farris Iman Leong Bin Abdullah, Dr., Universiti Sains Malaysia
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: MFLeong
Record Dates: First submitted 2021-03-10; First posted 2021-03-16 (Actual); Last update posted 2025-09-10 (Actual); Status verified 2025-09

CONDITIONS: Cancer of Head and Neck
Keywords: Mindfulness; Posttraumatic Growth; Hope; Optimism; Quality of Life
MeSH Terms: conditions — Head and Neck Neoplasms | interventions — Mindfulness-Based Stress Reduction

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mindfulness-based Stress Reduction (MBSR) (Experimental): MBSR will be conducted in a group of 10 for each session. The MBSR modules covered over 8 sessions, 1 hour in each session. The sessions will be held every week according to the patient's appointment date for chemotherapy treatment.
  Interventions: Behavioral: Mindfulness-based Stress Reduction (MBSR)
- Control (No Intervention): The subjects in the TAU control group will be assigned for non-therapeutic sessions at the same time and of equal duration to that of the MBSR group

INTERVENTIONS:
Behavioral: Mindfulness-based Stress Reduction (MBSR) — The term 'mindfulness' refers to mindful awareness as a way of being - a knowing and experiencing of feelings, thoughts, and perceptions as they arise and pass away each moment. It is a way of relating to all experiences in an open, receptive way, without judging experiences as good or bad (grasping at them or pushing them away). Mindfulness employed two styles of meditations: concentrative meditation involves intentionally focusing attention on a chosen object (e.g. the sensations of breathing) in a sustained way, while receptive meditation involves monitoring the content of experience (e.g. sensations, emotions, thoughts, sounds, etc.) in a non-reactive and non-judgmental way, from moment to moment, with the goal being to recognize the nature of emotional and cognitive patterns. Mindfulness-based stress reduction (MBSR) is an 8-week, standardized group intervention consisting of mindfulness meditation and gentle yoga that is designed to have applications for stress, pain, and illness
  Arms: Mindfulness-based Stress Reduction (MBSR)

SUMMARY:
Head and neck cancer is a group of biologically similar cancers which cause deleterious impact, such as the complication of facial disfigurement which may increase the psychological vulnerability of patients due to the society's emphasis on physical attractiveness. The appearance of facial disfigurement can increase depression and reduced quality of life (QoL) in head and neck cancer patients. Among the positive psychology developed in cancer patients despite their negative experience of cancer and the adverse effects of its treatment are posttraumatic growth (PTG) and hope which may enhance the QoL of cancer patients. Several psychosocial interventions have been suggested to enhance positive psychology in cancer patients and increase in their QoL. Data is lacking on the efficacy of mindfulness-based stress reduction (MBSR) on enhancing positive psychology (such as PTG, optimism and hope) and QoL among head and neck cancer patients. This is a multicentre, 2-armed longitudinal double blind randomized control trial aimed to test the study hypotheses of:

1. Head and neck cancer patients in the mindfulness-based stress reduction (MBSR) group reported significantly increase in posttraumatic growth (PTG), hope, optimism, and quality of life compared with those in the control group at post-intervention and 12 weeks after completion of intervention when compared with pre-intervention.
2. PTG, hope and optimism exerts partial mediation effects on the relationship between MBSR and quality of life among head and neck cancer patients.

DETAILED DESCRIPTION:
As head and neck cancer differ from other types of cancer due to the complication of facial disfigurement which may increase the psychological vulnerability of patients due to the society's emphasis on physical attractiveness. Moreover, a number of devastating complications of the cancer itself and the side effects of its treatment such as fatigue, pain, problem with speech and swallowing, breathing problem, mucositis, xerostomia, and trismus which further exerts detrimental effects on many functions and activities of daily living which causes further psychological distress and decreasing quality of life. Hence, it is of utmost importance to investigate on psychosocial interventions which could enhance PTG, hope, optimism and QoL of head and neck cancer patients which in turn bring about the ultimate outcome of restoring mental and physical well-being of the cancer survivors. Mindfulness-based stress reduction (MBSR) have been reported to enhance positive psychology in cancer patients. But the effect of MBSR on PTG, hope, optimism, and QoL among head and neck cancer patients have not been studied. Hence, there is a need to conduct a 2-armed randomized control trial to evaluate the effects of MBSR on PTG, hope, optimism, and QoL compared with control group with treatment-as-usual (TAU) across time.

Below are the objectives of this study:

General objective:

To examine the effects of mindfulness-based stress reduction (MBSR) on posttraumatic growth (PTG), hope, optimism, and quality of life among head and neck cancer patients.

Specific objectives:

1. To examine the changes in the degree of posttraumatic growth (PTG), hope, optimism, and quality of life of head and neck cancer patients in the MBSR group compared with those in the TAU control group at post-intervention and 12 weeks after intervention compared with pre-intervention.
2. To evaluate the mediation effects of PTG, hope and optimism on the relationship between MBSR and quality of life among head and neck cancer patients.

Study Setting:

The study will be conducted the Oncology and Otorhinolaryngology unit of Advanced Medical and Dental Institute, Universiti Sains Malaysia and Oncology and Otorhinolaryngology unit of Universiti Kebangsaan Malaysia Medical Centre. The Oncological and Otorhinolaryngology units of AMDI, USM have about 200-250 registered head and neck cancer patients currently under follow up. These units receive new cases of head and neck cancer every week. While the Department of Otorhinolaryngology and Department of Oncology of UKMMC have an estimated 350-400 registered head and neck cancer patients while the Department of Oral and Maxillofacial Surgery of UKMMC has an estimated 100-150 registered oral cancer patients under follow up (oral cancer is grouped under head and neck cancer).

Study design:

This is a multicentre, 2-armed longitudinal double blind randomized control trial which is expected to run for a duration of 2 years.

Sample size:

The sample size is determined based on G-Power 3.1.9.2 for repeated measures, between-within interaction ANOVA. Based on the previous study Lengacher et al (2009), the sample size was calculated based on the medium effect size (0.41), an alpha of 0.05, study power of 0.8 and it is two-tailed. In anticipation of a drop-out rate of 20%, the estimation for sample size is 110 respondents for total respondents and 55 respondents for each group.

Sampling method:

Sampling method use in this study is by consecutive sampling.

Recruitment of subjects:

The participants were recruited from the source population which included all newly diagnosed head and neck cancer patients who has been treated only with surgery or still remain untreated registered under the Oncology and Otorhinolaryngology unit of Advanced Medical and Dental Institute, Universiti Sains Malaysia and Oncology and Otorhinolaryngology unit of Universiti Kebangsaan Malaysia Medical Centre. These patients will be approached by the research team and explained on the study objectives and procedures.

Randomization:

Participants will be randomized into two groups, such as mindfulness-based stress reduction (MBSR) group and TAU control group. The participants will be randomized into one of the three groups in a 1:1 allocation ratio by block randomization. The allocation sequence is concealed in a sealed, opaque, sequential numbered envelope.

Data collection:

Data collection is carried out by a research assistant who is not involved in conduct of the study and data analysis. In the pre-intervention phase (T1), the participants in the two groups are administered the following questionnaires:

(i) Socio-demographic and clinical questionnaire which includes age, gender, marital status, monthly income, stage of cancer and type of head and neck cancer.

(ii) The Posttraumatic Growth Inventory-Short Form (PTGI-SF) to assess the degree of PTG of the participants (iii) The Dispositional Hope Scale to assess the degree of hope of the participants (iv) The Life Orientation Test-Revised (LOT-R) to assess the degree of optimism (v) The Functional Assessment of Cancer Therapy - Head & Neck (FACT-H & N) to assess the degree of quality of life

Then the assessments with the following questionnaires are repeated immediately post-intervention (T2) and 12 weeks after intervention (T3) among participants in all the two groups:

(i) The Posttraumatic Growth Inventory-Short Form (PTGI-SF) to assess the degree of PTG of the participants (ii) The Dispositional Hope Scale to assess the degree of hope of the participants (iii) The Life Orientation Test-Revised (LOT-R) to assess the degree of optimism (iv) The Functional Assessment of Cancer Therapy - Head & Neck (FACT-H & N) to assess the degree of quality of life

Blinding:

The participants will be blinded for the study as randomization into designated groups are conducted by a research assistant not involved in the study and the allocation is concealed in opaque, sequential numbered envelope. Therefore, the participants will not know which group they are allocated to. Although participants in the MBSR group undergo psychosocial intervention earlier, the participants in the control group (who are assigned TAU) will also undergo non-therapeutic sessions with the same time and duration as that of the MBSR group.

The researchers will be blinded for the study as randomization of participants into designated groups are conducted by a research assistant not involved in the conducting the study and data analysis. Data collection will also be caried out by the research assistant who is not involved in conducting the study and data analysis and blinded regarding the hypotheses of the study. Moreover, the data analysis will be performed out by statisticians who are not involved in conducting the study and blinded regarding the hypotheses of the study.

Interventions:

The MBSR intervention will be conducted in a group of 10 for each session. The ACT and MBSR modules covered over 6 sessions, 2.5 hours in each session. The sessions will be held every week according to the patient's appointment date for chemotherapy treatment.

Therapists:

The trainee therapists are four post-graduate students who enrolled in their Doctor of Philosophy (Ph.D.) in psychology. They received training approximately 16 hours of MBSR intervention. In the MBSR training, the trainee therapists will learn the basic overview and concepts of MBSR including mindfulness, body scan and yoga. Besides, they also will experiential learning about formal and informal practices, recording and home practices.

Data analysis:

Data analysis will be performed using SPSS version 26 software. Descriptive statistics will be used to analyze demographic data while inference analyses will be used to evaluate the significant difference between intervention and waitlist groups. In order to identify the efficacy of mindfulness-based stress reduction (MBSR) on the measured variables, several tests will be carried out. The comparison of mean differences pre-intervention (T1), post-treatment (T2) and 12 weeks after intervention (T3) will be examined to determine whether any changes in the measured variables (PTG, hope, optimism, QoL) in the MBSR and control groups across the three timelines by using mixed linear model. The effect sizes will be calculated to determine how substantially patients' perception towards measured variables changed with and without MBSR interventions. Statistical significance is set at p < 0.05 and two-tailed.

ELIGIBILITY:
Inclusion criteria:

* Those who are newly diagnosed with head and neck cancer confirmed by histopathological examination report at any stage of cancer and who already completed surgical treatment and currently undergoing adjuvant treatment (such as chemotherapy and/or radiotherapy/brachytherapy or immunotherapy)

  . Those who are literate in the Malay language (Bahasa Melayu)
* Age 18 years and above.

Exclusion criteria:

* Those with history of pre-existing psychiatric illnesses, such as depression, anxiety disorders, schizophrenia, schizophreniform disorder, schizoaffective disorder, delusional disorder, brief psychotic disorder, bipolar mood disorder, posttraumatic stress disorder, obsessive compulsive disorder, and neurodevelopmental disorders (patients are screened with Mini International Neuropsychiatric Interview to exclude these disorders).
* Those with history of illicit drug intake and those with substance use disorder, alcohol use disorder, substance-related disorders and alcohol-related disorders (patients are screened with urine dipstick for drugs and Mini International Neuropsychiatric Interview to exclude these conditions).
* Those with history of medical illnesses which can induced psychiatric symptoms such as stroke, coronary heart disease, congestive cardiac failure, COPD, bronchial asthma, systemic lupus erythematosus, rheumatoid arthritis, renal failure, hepatic failure, endocrine disorders, multiple sclerosis, Parkinson's Disease, and epilepsy.
* Those who are currently on any psychotherapy or counselling sessions.
* Those who are physically unfit to perform intervention.
* Those who exhibit cognitive impairment (patients are screen with Montreal Cognitive Assessment, in which those with score of < 25/30 will be excluded)

  * Those with suicidal tendency
  * Those who are pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2023-06-30 (Actual)

PRIMARY OUTCOMES:
Change in quality of life of head and neck cancer patients at 6 weeks immediately after completion of intervention and 12 weeks after completion of intervention | pre-intervention, 6 weeks- immediately after completion of intervention, and 12 weeks after completion of intervention
  Functional Assessment of Cancer Therapy - Head & Neck (FACT-H & N) is a self-reported tool which measures quality of life in patients with head and neck cancer. FACT-HN consists of 39 items and consists of 5 subscales: physical well-being (7 items), social/family well-being (7 items), emotional well-being (6 items), functional well-being (7 items) and head & neck cancer additional concerns (12 items). Each item is scored in a 5-point Likert scale ranging from 0= Not at all to 4= Very much. Hence, the total score range from 0 to 156. The higher the score, the greater is the degree of QoL. The tool also registered excellent psychometric properties. The FACT-H & N has been translated and validated in the Malaysian cancer population. All the subscales have moderate to good internal consistency with Cronbach's α ranging from 0.65 to 0.87. In this study, it is used to assess level of QoL among the participants.

SECONDARY OUTCOMES:
Change in level of hope of head and neck cancer patients at 6 weeks immediately after completion of intervention and 12 weeks after completion of intervention | pre-intervention, 6 weeks- immediately after completion of intervention, and 12 weeks after completion of intervention
  Dispositional Hope Scale is a self-rated 12 items scale which assesses the responder's level of hope. It comprised of 2 subscales which incorporates Snyder's cognitive model of hope i.e. (a) Agency (goal-directed energy) and (b) Pathways (planning to accomplish goals). 4 of the 12 items assess agency while another 4 items assess pathways. The other 4 items are fillers. Each item is scored using Likert-point scale from 1= Definitely False to 4= Definitely True. Hence, the total score range from 8 to 32. The higher the total score, the greater is the degree of hope. The Malay version of Hope Scale demonstrated Cronbach's alpha of 0.716. Intraclass correlation coefficient (ICC) gave a good score of 0.67 (95% CI: 0.57-0.75). Confirmatory factor analysis demonstrated 2 factors in which there are 4 items for each factor as in the original version of Hope Scale. In this study, it is used to assess level of hope among the participants.
Change in optimism of head and neck cancer patients at 6 weeks immediately after completion of intervention and 12 weeks after completion of intervention | pre-intervention, 6 weeks- immediately after completion of intervention, and 12 weeks after completion of intervention
  The Life Orientation Test-Revised (LOT-R) has 6 coded items with 3 framed in each direction, which are optimism and pessimism. The revision omitted or rewrote items that did not focus on explicit expectations. It has good internal consistency and stable over time. The positive and negative subsets are more strongly related to each other than those in the original Life Orientation Test. Each item is scored in a Likert scale range from 0 to 4. The total score range from 0 to 24. The higher the total score, the greater is the degree of optimism. The Malay version of LOT-R demonstrated intraclass correlation coefficient (ICC) gave a good score of 0.62 (95% CI: 0.50-0.71). Confirmatory factor analysis demonstrated 2 factors in which there are 3 items for each factor as in the original version of LOT-R with factor loading ranging from 0.46 to 0.72. In this study, it is used to assess the level of optimism of the participants.
Change in posttraumatic growth of head and neck cancer patients at 6 weeks immediately after completion of intervention and 12 weeks after completion of intervention | pre-intervention, 6 weeks-immediately after completion of intervention, 12 weeks after completion of intervention
  Posttraumatic Growth Inventory-Short Form (PTGI-SF) is the shorter version of the original Posttraumatic Growth Inventory and consists of 10 items where each of the 5 factors in posttraumatic growth is measured by 2 items. The higher the PTGI-SF score, the higher the level of posttraumatic growth in the individual being assessed. PTGI could be substituted by PTGI-SF with little loss of information. Each item is scored in a Likert scale from 0 to 4. Hence, the total score range from 0 to 50. The higher the total score, the greater the degree of posttraumatic growth. The PTGI-SF Malay version has good internal consistency which demonstrated Cronbach's alpha of 0.887 with the Cronbach's alpha of the 5 factors ranging from 0.700 to 0.813. Intraclass correlation coefficient (ICC) gave a good score of 0.75 (95% CI: 0.67-0.81). In this study, it is used to assess level of posttraumatic growth among the participants.

CONTACTS AND LOCATIONS:
Overall Officials: Mohammad Farris Iman Leong Bin Abdullah, Dr Psych, Principal Investigator — Advanced Medical and Dental Institute, Universiti Sains Malaysia
Locations (1):
- Advanced Medical and Dental Institute, Universiti Sains Malaysia, Kepala Batas, Pulau Pinang, Malaysia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Zhang Z, Zhang Q, Lu P, Shari NI, Nik Jaafar NR, Mohamad Yunus MR, Leong Bin Abdullah MFI. MBSR effects on positive psychological traits and experiential avoidance in head and neck cancer: a randomized controlled trial. Eur J Psychotraumatol. 2025 Dec;16(1):2501822. doi: 10.1080/20008066.2025.2501822. Epub 2025 May 19. PMID 40387873
- [Derived] Zhang Z, Leong Bin Abdullah MFI, Shari NI, Lu P. Acceptance and commitment therapy versus mindfulness-based stress reduction for newly diagnosed head and neck cancer patients: A randomized controlled trial assessing efficacy for positive psychology, depression, anxiety, and quality of life. PLoS One. 2022 May 10;17(5):e0267887. doi: 10.1371/journal.pone.0267887. eCollection 2022. PMID 35536828